CLINICAL TRIAL: NCT03568422
Title: A Phase Ib and Open Label Phase II Study of CFI-402257 in Combination With Weekly Paclitaxel in Patients With Advanced/Metastatic HER2-Negative Breast Cancer
Brief Title: CFI-402257 in Combination With Paclitaxel in Patients With Advanced/Metastatic HER2-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Stand Up To Cancer (Other); Canadian Breast Cancer Foundation (Other); Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I236
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CFI-402257; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CFI-402257 + Paclitaxel (Experimental): Oral CFI-402257 on intermittent schedule:* days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
  Interventions: Drug: CFI-402257; Drug: Paclitaxel

INTERVENTIONS:
Drug: CFI-402257 — Orally taken on intermittent schedule (days 1, 2, 8, 9, 15 & 16
Drug: Paclitaxel — 80 mg/m2 IV days 1, 8 & 15 every 28 days

SUMMARY:
The standard or usual treatment for this disease is to undergo chemotherapy to slow the spread of disease and relieve some symptoms of cancer. One of the standard types of chemotherapy is a drug called paclitaxel (Taxol) given in a low dose every week for three out of four weeks.

CFI-402257 is a new type of drug for breast cancer. Laboratory tests show that it may help slow the growth of breast cancer. This drug has been shown to shrink tumours in animals. CFI-402257 has been studied in a few people and appears well tolerated with little side effects. CFI-402257 seems promising but it is not clear if it can offer better results when given with paclitaxel compared to paclitaxel alone.

DETAILED DESCRIPTION:
Phase I:

The purpose of the first phase of the study is to find the highest dose of CFI-402257 that can be tolerated without causing very severe side effects when receiving paclitaxel. This is done by starting at a dose lower than the one that is tolerated in patients when given on its own. Participants are given CFI-402257 together with paclitaxel and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then new participants will be given a higher dose of CFI-402257. Participants joining this study later on will get higher doses of CFI-402257 than participants who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

Phase II:

The purpose of the second phase will be to find out the effect that CFI-402257 has on breast cancer, using doses found to be safe in the first phase of the study, when given with paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed diagnosis of breast cancer that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists, and for which systemic therapy is indicated. Only female patients will be enrolled
* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block. Biopsies are optional but strongly encouraged for patients with accessible disease suitable for biopsy. The timing of tumour biopsies for patients who provide informed consent and are willing is prior to treatment (after enrollment) and again no later than the end of the day following the day 8 paclitaxel infusion. Lesions planned for biopsy may not be the only target lesion.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 21 days prior to enrollment (within 28 days if negative). For phase Ib, patients are not required to have measurable disease as defined by RECIST 1.1 but must not have bone-only or marker only disease. For phase II, all patients must have measurable disease as defined by RECIST 1.1. The criteria for defining measurable disease are as follows:

Chest xray ≥ 20mm; CT scan ≥ 10mm (longest diameter); Physical exam ≥10mm; Lymph nodes by CT scan ≥ 15mm (measured in short axis)

* Patients must be ≥18 years of age.
* Patients must have an ECOG performance status of 0 or 1.
* Patients must be able to swallow oral medications
* Patients must have received at least one non-taxane containing chemotherapy regimen for advanced or metastatic disease unless:

  1. they have relapsed within 6 months of completion of adjuvant/neoadjuvant chemotherapy and the regiment did not contain taxane, or,
  2. they have received taxane and/or anthracycline-containing adjuvant/neoadjuvant chemotherapy 6 or more months prior to relapse or;
  3. they have a documented contraindication to palliative chemotherapy other than weekly paclitaxel.
* Patients must not be considered appropriate for endocrine therapy and must not have received taxanes in the metastatic setting.
* Patients may have received other therapies including endocrine therapy, immunotherapy, and/or targeted therapies (including CDK4/6 inhibitors).
* Patient may NOT have had previous exposure to any therapy within the pharmacological class (TTK/MPS1 inhibitor).
* Patients must have recovered (to at least grade 0 or 1) from all reversible toxicity other than alopecia related to prior chemotherapy or systemic therapy and have adequate washout as follows:
* Longest of one of the following:

  * Two weeks,
  * 5 half-lives for investigational agents,
  * Standard cycle length of standard therapies (e.g. at least 3 weeks for capecitabine.
* Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of enrollment. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG.
* Previous surgery is permitted provided that a minimum of 21 days (3 weeks) have elapsed between any major surgery and date of enrollment, and wound healing has occurred.
* Absolute neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥100 x 10^9/L
* Bilirubin ≤ 1.0 x ULN
* AST and ALT ≤3.0 x ULN and ≤ 5.0 x ULN (if patient has liver mets)
* Serum creatinine ≤ 1.5 x ULN or
* Creatinine clearance ≥ 60mL/min
* Women of childbearing potential must have agreed to use a highly effective contraceptive method
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.

Exclusion Criteria:

* Patients with a history of other untreated malignancies or malignancies which required therapy within the past 2 years. Patients with other malignancies of a nature that do not require treatment may be eligible after consultation with the CCTG.
* Patients with HER2 positive breast cancer.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should ahve a LVEF ≥ 50%
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with history of central nervous system metastases or spinal cord compression unless have received definitive treatment, are clinically stable and do not require corticosteroids.
* Patients who have contraindications to treatment with paclitaxel and/or neuropathy > grade 1.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Pregnant or breastfeeding women.
* Prohibited medications as listed in Appendix V Table 1
* Patients treated with full-dose warfarin. Patients with history of deep vein thrombosis or pulmonary embolus who are being treated with therapeutic doses of low molecular weight heparin, direct factor Xa inhibitors or prophylactic dose anticoagulants may be enrolled.
* Patients with a medical condition that could impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, Study Chair — Princess Margaret Cancer Centre, Toronto, ON; Mihaela Mates, Study Chair — Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, ON
Locations (4):
- Canada (4):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were five dose levels in the phase I component of this study with respectively 4, 3, 6, 7, and 6 patients enrolled. Based on the results from patients on dose levels 4 and 5, dose level 3 was expanded with 11 additional patients enrolled. From the results of a total of 17 patients enrolled in this dose level, dose level 3 was declared as the recommended phase II dose and all 17 patients enrolled in dose level 3 were considered to be Phase II patients for the analyses.
Groups:
- Phase I: Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 84 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase 1: Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 112 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase 1: Dose Level 3 (CFI-402257 168 mg + Paclitaxel 80 mg/m2); Expansion Cohort: CFI-402257 168 mg + Paclitaxel 80 mg/m2: Oral CFI-402257 168 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I: Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)): Oral CFI-402257 210 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I: Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 252 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2) | Phase 1: Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2) | Phase 1: Dose Level 3 (CFI-402257 168 mg + Paclitaxel 80 mg/m2) | Phase I: Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)) | Phase I: Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2) | Expansion Cohort: CFI-402257 168 mg + Paclitaxel 80 mg/m2
Started | 4 | 3 | 6 | 7 | 6 | 11
Completed | 4 | 3 | 6 | 7 | 6 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the study
Groups:
- Phase 1 Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 84 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 112 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 168 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)): Oral CFI-402257 210 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Phase I Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 252 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)) | Phase I Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2) | Total
Number analyzed (Participants) | 4 | 3 | 17 | 7 | 6 | 37
Age, Continuous [Median (Full Range); unit: years] | 58 [30 to 59] | 48 [47 to 51] | 58 [40 to 72] | 62 [46 to 70] | 65 [50 to 72] | 59 [30 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 17 | 7 | 6 | 37
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 2 | 12 | 6 | 5 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 17 | 7 | 6 | 37
ECOG (Eastern Cooperative Oncology Group) Performance Status [Count of Participants; unit: Participants] — grade 0: fully active, able to carry on all pre-disease performance without restriction; grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; grade 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; grade 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours; grade 4: completely disabled, cannot carry on any self-care, totally confined to bed or chair; grade 5: dead.
  Participants
    0 | 3 | 2 | 5 | 5 | 4 | 19
    1 | 1 | 1 | 12 | 2 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose for CFI-402257
Description: The maximum tolerated dose of CFI-402257 for phase II study identified by a standard 3+3 design to escalate the dose of CFI-402257.
Time Frame: During cycle 1 (28 days)
Population: There were five dose levels in the phase I component of this study with respectively 4, 3, 6, 7, and 6 patients enrolled. Based on the results, dose level 3 was declared as the recommended phase II dose.
Measure: Number; unit: mg
Groups:
- CFI-402257 + Paclitaxel: Oral CFI-402257 at 5 dose levels on intermittent schedule:
  days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
Arm/Group | CFI-402257 + Paclitaxel
Number analyzed (Participants) | 26
mg | 168

2. Primary Outcome: Phase II: Overall Response Rate Using RECIST 1.1
Description: Percentage of patients with a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: Participants who received Dose Level 3 in Phase I and in the expansion cohort are combined for analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 168 mg on intermittent schedule:* days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
Arm/Group | Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2)
Number analyzed (Participants) | 17
Participants | 1

3. Secondary Outcome: Phase II: Clinical Benefit Rate Determined by Complete Response, Partial Response or Stable Disease
Description: Percentage of patients with a complete response (CR) or partial response (PR), or with stable disease (SD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), <30% decrease in the sum of the longest diameter of target lesions but <20% increase in the sum of the longest diameter of target lesions>16 weeks of duration; Overall clinical benefit = CR + PR+SD.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level 3 and Expansion Cohort ( CFI-402257 168 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 168 mg on intermittent schedule:* days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
Arm/Group | Phase I Dose Level 3 and Expansion Cohort ( CFI-402257 168 mg + Paclitaxel 80 mg/m2)
Number analyzed (Participants) | 17
Participants | 8

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Phase I Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2): Oral CFI-402257 84 mg on intermittent schedule: days 1, 2, 8, 9, 15 & 16 q4w Plus Paclitaxel 80 mg/m2 IV days 1, 8 & 15 every 28 days
Arm/Group | Phase I Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2) | Phase I Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)) | Phase I Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2)
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/3 | 16/17 | 5/7 | 4/6
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 3/17 | 2/7 | 1/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 17/17 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2) (N=4) | Phase I Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2) (N=3) | Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2) (N=17) | Phase I Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)) (N=7) | Phase I Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2) (N=6)
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Other metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (CFI-402257 84 mg + Paclitaxel 80 mg/m2) (N=4) | Phase I Dose Level 2 (CFI-402257 112 mg + Paclitaxel 80 mg/m2) (N=3) | Phase I Dose Level 3 and Expansion Cohort (CFI-402257 168 mg + Paclitaxel 80 mg/m2) (N=17) | Phase I Dose Level 4 (CFI-402257 210 mg + Paclitaxel 80 mg/m2)) (N=7) | Phase I Dose Level 5 (CFI-402257 252 mg + Paclitaxel 80 mg/m2) (N=6)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 12 | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 10 | 4 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 8 | 1 | 2
Fatigue (General disorders) | 4 | 1 | 13 | 6 | 6
Non-cardiac chest pain (General disorders) | 2 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 5 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 9 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 3 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 7 | 4 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 6 | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0 | 1 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 10 | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 9 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 0
Other eye disorders - Double vision (Eye disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 12 | 2 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Other infections and infestations - Common cold (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6 | 2 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 13 | 3 | 4
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0
Other skin and subcutaneous tissue disorders - Thinning of eyebrows and eyelashes, and Erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 1 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 1 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 2 | 1 | 1
Fever (General disorders) | 0 | 1 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 2 | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 0 | 0
Other surgical and medical procedures - Back pain due to biopsy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 2 | 0 | 0
Other eye disorders - Stye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Belching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0 | 0
Other general disorders, administration site conditions - Pain to site of PleurX (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Shingles (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Other infections and infestations - COVID-19 infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Other musculoskeletal and connective tissue disorder - Port site pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Other neoplasms benign, malignant and unspecified - Lump on right neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Other renal and urinary disorders - Intermittent delay in starting urination (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Other respiratory, thoracic and mediastinal disorders - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Other skin and subcutaneous tissue disorders - Erythema around Port-a-Cath, Skin discolouration, and (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Other vascular disorders - Small non-occlusive thrombosis in bilateral gonadal veins (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Other infections and infestations - Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vaginismus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT03568422/Prot_SAP_000.pdf